CLINICAL TRIAL: NCT06646874
Title: Active Video Game Using Virtual Reality Influence Cognitive Ability in Sedentary Female University Students: Randomized Clinical Trial
Brief Title: Active Video Game Influence Cognitive Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RHPT/023/007
Record Dates: First submitted 2024-08-19; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Physical Inactivity
Keywords: Virtual Reality; Cognitive performance; Physical activity; Sedentary female student
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were required to attend one experimental session in a random order using Microsoft Excel's (Microsoft Corp., Redmond, WA, USA) random list function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group completed the MoCA pre- and post-tests 20 minutes apart. A debriefing was conducted for the participants following the conclusion of the experiment.
- VR group (Experimental): Each participant in the VR group completed a five-minute familiarization session with the VR game before the experimental session. Following the familiarization session, participants in the VR group were instructed to complete the Montreal Cognitive Assessment (MoCA) Arabic version (pre-test: Arabic version 8.1 and post-test: Arabic version 8.2)
  Interventions: Behavioral: VR game

INTERVENTIONS:
Behavioral: VR game — Each participant in the VR group completed a five-minute familiarization session with the VR game before the experimental session. Following the familiarization session, participants in the VR group were instructed to complete the Montreal Cognitive Assessment (MoCA) Arabic version (pre-test: Arabic version 8.1 and post-test: Arabic version 8.2)
  Arms: VR group

SUMMARY:
The experiment was conducted at the Human Biomechanics Laboratory of the College of Applied Medical Sciences of Prince Sattam bin Abdulaziz University between February 2024 and May 2024. During the briefing, all questions were answered to ensure that participants understood the experiment and its objectives. On the day of the experiment, demographic information was collected, including age, height, weight, body mass index (BMI), and preferred leg. An Eye-Level Weight Beam scale (Detecto, Webb City, MO, USA) was used to determine the weight and height of the subjects. To identify the preferred leg, participants were observed ascending stairs or kicking a ball.

Participants were recruited and assigned to one of two groups, either the control group or the VR group. Participants were required to attend one experimental session in a random order using Microsoft Excel's (Microsoft Corp., Redmond, WA, USA) random list function. The VR group was required to play a 20-minute game of Beat Saber VR, while the control group was asked to sit quietly for 20 minutes without any activities assigned. This study used an accelerometer from ActivPal (PAL Technologies Ltd, Glasgow, UK) to capture the PA levels of the VR group throughout the VR game. Following previously published validation studies and manufacturer recommendations, a strip of Tegaderm (3M, St. Paul, MN) was attached to the preferred leg's front thigh.

ELIGIBILITY:
Inclusion Criteria:

* Female college students
* Low physical activity (inactive)
* Age (18 to 23 years)
* No previous medical condition affecting PA level
* No visual impairments
* Have never experienced the VR game used in the trial

Exclusion Criteria:

* Male students
* Physically active

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 20 minutes
  Developed as a screening instrument to detect mild cognitive impairment, the Montreal Cognitive Assessment (MoCA) uses a series of questions to assess cognitive impairment. A paper-and-pencil assessment is administered and scored out of 30 points. In addition to attention, concentration, executive functions, memory, language, visuospatial skills, abstraction, calculation, and orientation, the MoCA assesses several cognitive domains. There are 56 languages and dialects translation of the MoCA and it is widely used throughout the world
ActivPal | 20 minutes
  The ActivPAL is a posture and activity tracker that uses a tri-axial accelerometer to measure movement and activity. The device collects information such as bouts of sitting, lying, standing, and stepping, and allows data to be retrieved by week, day, or hour. As a valid and reliable tool to detect PA, ActivPal can be used in a variety of populations and settings (64). From the ActivPal, the following variables were collected for each participant in the VR group: total MET, total number of steps, total time stepping, number of sit-to-stands, and number of stands-to-sit.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Biomechanics Laboratory of the College of Applied Medical Sciences of Prince Sattam bin Abdulaziz University, Al Kharj, Central, Saudi Arabia